CLINICAL TRIAL: NCT03563703
Title: Transfer of Technological Innovations to Nursing Practice: A Contribution to the Prevention of Infections
Acronym: TecPrevInf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other); Associação Portuguesa de Acessos Vasculares (Unknown); Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Responsible Party: Principal Investigator, Anabela Salgueiro-Oliveira, Ph.D, Assistant Professor, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TecPrevInf
Record Dates: First submitted 2018-05-09; First posted 2018-06-20 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Catheterization, Peripheral
Keywords: Catheterization, Peripheral; Ultrasound; Near Infrared Light
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Once eligibility, informed consent and assent are confirmed, participants will be randomly assigned, in the appropriate age stratum, to 1 of 2 groups: peripheral intravenous catheterization with the standard approach or with the help of either ultrasound or near-infrared vascular imaging. Randomization will be achieved with the use of an online, computer-generated program.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Because of the physical nature of the interventions, it will not be possible to conceal the group allocation from the nurses or trial participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound imaging (Experimental): Ultrasonography offers visual information about the size and depth of blood vessels, potentially facilitating intravenous placement of the needle in real time.
  Interventions: Device: Ultrasound
- Near-infrared imaging (Experimental): Near-infrared imaging devices project near-infrared light onto the skin, which is absorbed by deoxygenated hemoglobin. The invisible image of the underlying vascular pattern is captured by the device, processed and projected, in real time, back onto the patient's skin using visible green light. This technology allows hands-free visualization of a vascular map to guide catheter placement.
  Interventions: Device: Near Infrared Light

INTERVENTIONS:
Device: Ultrasound — Ultrasound allows viewing veins and surrounding anatomical structures, making it easier to perform the placement of a cannula into a peripherally located vein in real time. This process allows the cannulation of veins that are unable to be visualised or palpated.
  Arms: Ultrasound imaging
Device: Near Infrared Light — Infrared technologies allows illuminating the vein with a near-infrared light, which is absorbed by blood and reflected by adjacent tissue.
  Arms: Near-infrared imaging

SUMMARY:
The insertion of peripheral vascular catheters (PVCs) is the most often invasive procedure performed in hospital settings. During hospitalization, the majority of patients need to have a PVC inserted. These devices are not risk-free, affecting patients' safety and well-being. In clinical settings, health professionals must deal with difficult venous accesses due to the patient's age, physical characteristics, clinical status, and medication, which hinder the PVC insertion. When veins are not visible or palpable, this may lead to successive puncture attempts, causing pain to the patient and discomfort to the nurse, which results in increased costs.

Guidelines state that puncture should be attempted only twice per professional, to a maximum of four attempts; against this recommendation and due to the patient's therapeutic needs and clinical situation, health professionals attempt to puncture multiple times in a single scenario. In this regard, health professionals should consider using specific technologies that help to select the vein and reduce the number of puncture attempts and catheter-related mechanical complications. Taking into account the multiplicity of existing technologies in the international market that assist health professionals in peripheral venous catheterization, ultrasound and infrared devices emerge in the literature as two of the most commonly used during this procedure.

These technologies were developed with the purpose of improving peripheral intravenous catheterization success rate and thus reducing the number and extent of the negative effects of multiple or unsuccessful attempts, with the additional purpose of avoiding the frustrations of health professionals in these scenarios. However, such technologies are still underused in clinical practice, since health professionals are not familiar with the use of these devices. Moreover, the costs associated with their purchase and maintenance may be considered as excessive in relation to the traditional method.

The project investigators aim to determine whether the use of either ultrasound or near-infrared vascular imaging will significantly improve the success rate of peripheral intravenous catheterization in adults on first attempt by nurses compared with the standard approach, reduce immediate related complications and improve patient and provider satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Participants who require peripheral intravenous catheterization as part of routine care;
* Participants whose primary nurse agrees to participate in the study;
* Participants who are able to give written assent or oral assent.

Exclusion Criteria:

* Confused and/or disoriented participants;
* Participants who are unable to communicate orally and/or in writing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Successful intravenous catheterization on the first attempt | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months., assessed up to 6 months
  Successful attempt is defined through the clear flush of the catheter with 5 mL of normal saline without extravasation.

SECONDARY OUTCOMES:
Number of attempts to successful intravenous catheter placement | Immediately following intervention, an average of 5 minutes. This outcome will be assessed through study completion, an average of 6 months.
Time to successful placement (in minutes) | From time of randomization until the time of successful intravenous catheter placement, assessed through study completion, an average of 6 months.
Patient satisfaction | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months.
  Evaluated through a self-report scale where the participant identifies a set of indicators associated to their satisfaction with the intervention, when compared to previous experiences.
Nurse satisfaction | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months.
  Evaluated through a self-report scale where the nurse identifies a set of indicators associated to their satisfaction with the intervention, when compared to previous experiences.
Immediate Complications | This outcome will be assessed immediately following intervention, an average of 20 minutes. This outcome will be assessed through study completion, an average of 6 months.
  Evaluated through a self-report scale where the nurse identifies a set of indicators associated to the occurrence of immediate complications during the procedure (extravasation, puncture of proximal anatomical structures, hematoma, etc.).
Patient anxiety (State-Trait Anxiety Inventory) | Anxiety will be assessed about ten minutes before and ten minutes after the intervention. This outcome will be assessed through study completion, an average of 6 months.
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger, Gorsuch, Lushene, Vagg, & Jacobs, 1983). It can be used in clinical settings to diagnose anxiety. Form Y, its most popular version, has 20 items for assessing trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Salgueiro-Oliveira, Ph.D, Principal Investigator — Assistant Professor
Locations (1):
- Centro Hospitalar e Universitário de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Marsh N, Webster J, Mihala G, Rickard CM. Devices and dressings to secure peripheral venous catheters to prevent complications. Cochrane Database Syst Rev. 2015 Jun 12;2015(6):CD011070. doi: 10.1002/14651858.CD011070.pub2. PMID 26068958
- [Background] Grune F, Schrappe M, Basten J, Wenchel HM, Tual E, Stutzer H; Cologne Quality Control Network. Phlebitis rate and time kinetics of short peripheral intravenous catheters. Infection. 2004 Feb;32(1):30-2. doi: 10.1007/s15010-004-1037-4. PMID 15007740
- [Background] Pujol M, Hornero A, Saballs M, Argerich MJ, Verdaguer R, Cisnal M, Pena C, Ariza J, Gudiol F. Clinical epidemiology and outcomes of peripheral venous catheter-related bloodstream infections at a university-affiliated hospital. J Hosp Infect. 2007 Sep;67(1):22-9. doi: 10.1016/j.jhin.2007.06.017. Epub 2007 Aug 27. PMID 17719678
- [Background] Abolfotouh MA, Salam M, Bani-Mustafa A, White D, Balkhy HH. Prospective study of incidence and predictors of peripheral intravenous catheter-induced complications. Ther Clin Risk Manag. 2014 Dec 8;10:993-1001. doi: 10.2147/TCRM.S74685. eCollection 2014. PMID 25525365
- [Background] Cicolini G, Manzoli L, Simonetti V, Flacco ME, Comparcini D, Capasso L, Di Baldassarre A, Eltaji Elfarouki G. Phlebitis risk varies by peripheral venous catheter site and increases after 96 hours: a large multi-centre prospective study. J Adv Nurs. 2014 Nov;70(11):2539-49. doi: 10.1111/jan.12403. Epub 2014 Mar 31. PMID 24684163
- [Background] Dorniak-Wall T, Rudaks L, Solanki NS, Greenwood J. Safe and correct use of peripheral intravenous devices. ANZ J Surg. 2013 Oct;83(10):764-8. doi: 10.1111/j.1445-2197.2012.06281.x. Epub 2012 Oct 4. PMID 23035825
- [Background] Ismailoglu EG, Zaybak A, Akarca FK, Kiyan S. The effect of the use of ultrasound in the success of peripheral venous catheterisation. Int Emerg Nurs. 2015 Apr;23(2):89-93. doi: 10.1016/j.ienj.2014.07.010. Epub 2014 Aug 15. PMID 25175514
- [Background] Partovi-Deilami K, Nielsen JK, Moller AM, Nesheim SS, Jorgensen VL. Effect of Ultrasound-Guided Placement of Difficult-to-Place Peripheral Venous Catheters: A Prospective Study of a Training Program for Nurse Anesthetists. AANA J. 2016 Apr;84(2):86-92. PMID 27311149
- [Background] Park JM, Kim MJ, Yim HW, Lee WC, Jeong H, Kim NJ. Utility of near-infrared light devices for pediatric peripheral intravenous cannulation: a systematic review and meta-analysis. Eur J Pediatr. 2016 Dec;175(12):1975-1988. doi: 10.1007/s00431-016-2796-5. Epub 2016 Oct 26. PMID 27785562